CLINICAL TRIAL: NCT05134935
Title: Defocus Incorporated Multiple Segment (DIMS) Spectacle Lenses Versus Orthokeratology Lenses (OKL) for Slowing Myopia Progression In Children Aged 6-12 Years. A Non-inferiority Randomized Clinical Trial. The NISDO Study.
Brief Title: Defocus (DIMS) Spectacles Versus Ortho-K Lenses (OKL) for Slowing Myopia Progression in Children Aged 6-12 Years.
Acronym: NISDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NISDO
Record Dates: First submitted 2021-11-15; First posted 2021-11-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Eyeglasses

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OKL (Active Comparator)
  Interventions: Device: Orthokerathology lenses (OKL)
- DIMS (Experimental)
  Interventions: Device: Defocus Incorporated Multiple Segment (DIMS) Spectacles

INTERVENTIONS:
Device: Defocus Incorporated Multiple Segment (DIMS) Spectacles — 18 months of therapy.
  Other Names: Defocus (DIMS) Spectacles
  Arms: DIMS
Device: Orthokerathology lenses (OKL) — 18 months of therapy.
  Other Names: Night lenses
  Arms: OKL

SUMMARY:
The goal of this non-inferiority randomized clinical trial is to compare the myopia control efficacy of Ortho-K lenses (OKL) and Defocus (DIMS) spectacles in myopic children aged 6-12 years. The main question it aims to answer is:

- Is the DIMS spectacle lens not worse than the OKL after 18 months of therapy?

The participants are randomly assigned to either OKL or DIMS spectacles and followed during 18 months of therapy.

ELIGIBILITY:
Inclusion criteria:

- Myopic children aged 6 to 12 years: Myopia of the 6 to 8-year-olds (inclusive): -1.00 to -4.75 D spherical component and up to -2.50 D of regular astigmatism (both eyes).

Myopia of the 9 to 12-year-olds (inclusive): -2.00 to -4.75 D spherical component and up to -2.50 D of regular astigmatism (both eyes).

* Anisometropia ≤ 1.50 D cycloplegic spherical equivalent refractive error.
* Best corrected visual acuity at age 6 to 12 years (inclusive): 0.8 Snellen (equivalent to ≥ 3/5 letter on the 0.8 line = 78 ETDRS letters)

Exclusion criteria:

* Manifest or intermittent squint.
* Contraindications to the use of OKL comprising (not exhaustive): keratoconus, chronic allergic conjunctivitis and keratoconjunctivitis sicca.
* Previous eye surgery.
* Chronic eye disease demanding daily use of eye drops.
* Non-compliance to eye examinations (unstable fixation or anxiety towards contact lenses).
* Previous myopia control treatment.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2025-12-02 (Actual); Study Completion 2025-12-02 (Actual)

PRIMARY OUTCOMES:
Axial length growth of the eye | 18 months
  Length in mm is measured 18 months after therapy

SECONDARY OUTCOMES:
Overall eye length growth, defined as the sum of axial length and choroidal thickness | 18 months
  Length in mm is measured 18 months after therapy

OTHER OUTCOMES:
Choroidal thickness | During 18 months of therapy
  Thickness is measured in um
Pupil size | 6 months
  Length in mm is measured 6 months after therapy
Vision related quality of life using the questionnaire PREP2 | Prior to and 9 months after treatment initiation
  Range from "strongly disagree" to "strongly agree"

CONTACTS AND LOCATIONS:
Overall Officials: Lou-Ann Andersen, Principal Investigator — Vejle Hospital
Locations (1):
- The Ophthalmic department, Vejle Hospital, Vejle, Southern Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-11-24): https://cdn.clinicaltrials.gov/large-docs/35/NCT05134935/SAP_001.pdf